CLINICAL TRIAL: NCT00615901
Title: Pilot Study of Dose Dense Adjuvant CMF (Cyclophosphamide, Methotrexate, Fluorouracil) at 14 and 10-11 Day Intervals for Women With Early Stage Breast Cancer
Brief Title: Dose Dense Adjuvant CMF (Cyclophosphamide, Methotrexate, Fluorouracil) at 14 and 10-11 Day Intervals for Women With Early Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-133
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: cyclophosphamide; methotrexate; fluorouracil; PEG-filgrastim
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Methotrexate; Fluorouracil; pegfilgrastim

ARMS (1):
- 1 (Experimental): This is a pilot study using 8 cycles of CMF (cyclophosphamide 600 mg/m2, methotrexate 40 mg/m2, and fluorouracil 600 mg/m2), at 14 day intervals supported by PEG-filgrastim for a cohort of 38 patients. A safety analysis will then be performed.
  Interventions: Drug: cyclophosphamide, methotrexate, fluorouracil, PEG-filgrastim

INTERVENTIONS:
Drug: cyclophosphamide, methotrexate, fluorouracil, PEG-filgrastim — C (cyclophosphamide) 600 mg/m2 M (methotrexate) 40 mg/m2 F (fluorouracil) 600 mg/m2 P (PEG-filgrastim ) 6 mg. Eight doses of CMF q 14 days with PEG-filgrastim administered approximately 24 hours after chemotherapy. Day 14, is also considered day 1 of the next cycle.

SUMMARY:
CMF (cyclophosphamide, methotrexate, fluorouracil) is used to treat early stage breast cancer. The combination, of these three drugs, has been used for approximately 30 years in the treatment of breast cancer, and has been shown to be safe and effective. It is usually given every 3 weeks. Doctors believe, based on other breast cancer trials, that giving this type of chemotherapy in a shorter amount of time, every 2 weeks or sooner, instead of every 3 weeks, may be better. The purpose of this study is to test the safety of these drugs, given every 2 weeks or sooner, to treat breast cancer. Other breast cancer chemotherapy regimens have shown to be more beneficial when the drugs are given more frequently.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed adenocarcinoma of the breast confirmed at MSKCC within 3 months of enrollment. Patients with inflammatory breast cancer are not eligible for the study. Pathology will be assessed in the standard fashion. Results of HER-2/neu, estrogen receptor, and progesterone receptor are required for study entry.
* The patient cannot be Her-2/neu over-expressing either by immunohistochemistry or FISH as per hospital laboratory standard whether institutional or outside laboratory.
* Patients must be > than or equal to 18 years of age
* Patients must have a Karnofsky score of > than or equal to 80
* Patients may have received hormonal therapy for the purpose of chemoprevention but must be willing to discontinue at least 24 hours prior to enrollment and while participating in this trial.
* Patients will have completed their definitive breast surgery (mastectomy or breast conserving surgery)
* Patients must be ready to begin therapy within 84 days from the final surgical procedure required to treat their primary tumor
* Patients must be stage I-II
* Absolute neutrophil count (ANC) > than or equal to 1500/µL and platelet count > than or equal to 100,000/µL
* Total bilirubin must be < than or equal to 1.1 mg/dL or within normal institutional limits if outside MSKCC. Transaminases (SGOT/AST and/or SGPT/ALT) may be up to < than or equal to 92.5 U/L or < than or equal to 2.5 x institutional upper limit of normal (ULN) if alkaline phosphatase is < than or equal to ULN, or alkaline phosphatase may be up to 4 x ULN if transaminases are < than or equal to ULN.
* Serum creatinine must be within 0.6-1.3 mg/dL or within normal institutional limits if outside MSKCC.
* Patients must be willing to discontinue sex hormonal therapy e.g., birth control pills, ovarian hormonal replacement therapy, etc., prior to enrollment. Women of childbearing potential must be willing to consent to using effective contraception while on treatment and for a reasonable period thereafter.
* Patients must give written, informed consent indicating their understanding and willingness to participate in the study.
* Brachytherapy after lumpectomy is permitted.

Exclusion Criteria:

* Stage III-IV breast cancer
* Prior chemotherapy or radiation therapy is excluded except for brachytherapy.Radiation for patients on this protocol will be given, if indicated, after the completion of chemotherapy.
* Pregnant or lactating patients
* Patients with a concurrently active second malignancy, other than adequately treated non-melanoma skin cancers or in situ cervical cancer. Patients with other non-mammary malignancies must have been disease-free for at least five years.
* Patients with unstable angina, congestive heart failure, current use of digitalis, betablockers, or calcium blockers for therapy of congestive heart failure, arrhythmia requiring medical therapy, or with a history of a myocardial infarction within 12 months.
* Patients with a psychiatric illness that would prevent them from understanding the nature of the investigational therapy and complying with protocol requirements.
* Patients with concurrent medical conditions, which, in the judgment of the investigator, would make them inappropriate candidates for study enrollment
* Patients with active, unresolved infections
* Patients that have known sensitivity to E. coli derived proteins, PEG-filgrastim, filgrastim, or any component products.
* Patients must be Her 2/neu non-over-expressing.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Drullinsky, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Mercy, Rockville Centre, New York
  - Memoral Sloan-Kettering Cancer Center at Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A (CMF at 14 Day Intervals): This is a pilot study using 8 cycles of CMF (cyclophosphamide 600 mg/m2, methotrexate 40 mg/m2, and fluorouracil 600 mg/m2), at 14 day intervals supported by PEG-filgrastim.
  cyclophosphamide, methotrexate, fluorouracil, PEG-filgrastim: C (cyclophosphamide) 600 mg/m2 M (methotrexate) 40 mg/m2 F (fluorouracil) 600 mg/m2 P (PEG-filgrastim ) 6 mg. Eight doses of CMF q 14 days with PEG-filgrastim administered approximately 24 hours after chemotherapy. Day 14, is also considered day 1 of the next cycle.
Period: Overall Study
Arm/Group | Cohort A (CMF at 14 Day Intervals)
Started | 38
Completed | 29
Not Completed | 9
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 7

BASELINE CHARACTERISTICS:
Arm/Group | Cohort A (CMF at 14 Day Intervals)
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 52 [38 to 78]
Gender [Count of Participants; unit: Participants]
  Female | 38
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients Who Completed 8 Cycles.
Description: the study regimen is deemed feasible and tolerable for patients with ANC > 1.5 on day 1 of treatment for all 8 cycles and absence of grade 3 or higher non-hematologic toxicity, excluding alopecia, nausea/vomiting and bone pain We will also evaluate the total number of days needed to complete all 8 cycles.
Time Frame: 2 years
Measure: Number; unit: participants
Groups:
- Cohort A (CMF at 14 Day Intervals): This is a pilot study using 8 cycles of CMF (cyclophosphamide 600 mg/m2, methotrexate 40 mg/m2, and fluorouracil 600 mg/m2), at 14 day intervals supported by PEG-filgrastim for a cohort of 38 patients. A safety analysis will then be performed.
  cyclophosphamide, methotrexate, fluorouracil, PEG-filgrastim: C (cyclophosphamide) 600 mg/m2 M (methotrexate) 40 mg/m2 F (fluorouracil) 600 mg/m2 P (PEG-filgrastim ) 6 mg. Eight doses of CMF q 14 days with PEG-filgrastim administered approximately 24 hours after chemotherapy. Day 14, is also considered day 1 of the next cycle.
Arm/Group | Cohort A (CMF at 14 Day Intervals)
Number analyzed (Participants) | 29
participants | 29

ADVERSE EVENTS:
Arm/Group | Cohort A (CMF at 14 Day Intervals)
Serious Adverse Events (participants affected / at risk) | 2/38
Other Adverse Events (participants affected / at risk) | 19/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (CMF at 14 Day Intervals) (N=38)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0)
Skin infection (Infections and infestations) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (CMF at 14 Day Intervals) (N=38)
Constipation (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Headache (Nervous system disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes